CLINICAL TRIAL: NCT02470819
Title: A Two Arm Pilot Study Utilizing Molecular Profiling to Find Potential Targets and Influence Treatments for Patients With Metastatic Breast Cancer or Advanced Gynecological Malignancies
Brief Title: Genomic and Proteomic Profiling Targets Influenced Treatment in Metastatic Breast Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator elected to end the study
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMEM-2014-DOD001
Record Dates: First submitted 2015-06-09; First posted 2015-06-12 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Metastatic Breast Cancer; Breast Tumor; Advanced Gynecologic Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — DNA Fingerprinting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Targeted Therapy (Experimental): Those who will receive targeted therapy based on their genetic profiling
  Interventions: Genetic: Genetic profiling

INTERVENTIONS:
Genetic: Genetic profiling — genetic profiling

SUMMARY:
The primary objective is to examine the impact on progression-free survival of targeted therapy for breast cancer suggested by proteomic and genomic profiling.

DETAILED DESCRIPTION:
To explore the impact of targeted therapy for breast cancer suggested by proteomic and genomic profiling using RPMA, targeted resequencing, IHC analysis, WGS, RNA-seq, and Exome sequencing on progression-free survival. When a molecular target cannot be identified, the patient will be treated with a therapy selected on an empirical basis by the investigator/treating physician at the individual site and will be followed for survival status. Only available, FDA-approved agents will be used.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of >3 months
* Diagnosis of metastatic breast cancer or an advanced gynecological malignancy with measurable disease
* Age greater than or equal to 18 years
* ECOG performance status of 0-1
* Able to undergo two biopsies to obtain tissue with first biopsy required and second biopsy optional
* Have failed or unable to tolerate previous treatment regimen
* Adequate organ and bone marrow function as defined by ANC ≥ 1.5 x 109/L; Hgb 9 g/dL; platelets greater than 100 x 109/L; creatinine ≤ 1.5 mg/dL; bilirubin ≤ 2.5 x ULN; AST and ALT ≤ 2.5 x ULN (or ≤ 5 x ULN if due to underlying liver metastases); INR ≤ 1.5 x ULN (except in the case of anticoagulation therapy)

Exclusion Criteria:

* Metastatic lesions that are not accessible to biopsy
* Symptomatic CNS metastasis
* Previous history of another malignancy within 5 years of study entry
* Uncontrolled concurrent illness
* Known HIV, HBB, and/or HCV infection
* Pregnant or breast feeding or childbearing potential and not using adequate birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 4 months
  Progression-free survival will be defined as the interval between the first dose of therapy and the occurrence of disease progression (fatal or non-fatal). Disease status will be assessed every 7 +/- 1 week until progression or time of treatment discontinuation, whichever is later. If progression is not observed at the end of therapy, patients will be assessed every 3 months until progression or further anti-cancer therapy.

SECONDARY OUTCOMES:
Tumor assessment | 4 months
  Radiographic response will be evaluated according to RECIST 1.1 criteria in all patients with measurable disease. All sites of disease must be evaluated using the baseline assessment methods. Confirmatory assessment of complete response or partial response must be performed no less than 4 weeks after the initial documentation of response.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Leyland-Jones, MD, Principal Investigator — Avera McKennan
Locations (1):
- Avera Cancer Institute, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No